CLINICAL TRIAL: NCT00630214
Title: Phase 2 Study of Routine Oral Calcium and Vitamine D Supplements to Prevent Hypocalcemia After Total Thyroidectomy in Papillary Thyroid Carcinoma Patients
Brief Title: Prevention of Hypocalcemia in Patients Undergoing Total Thyroidectomy Plus Central Neck Dissection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Chungnam National University (Other)
Responsible Party: Jong-Lyel Roh, MD, PhD, Chungnam National University Hospital & Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2004-03-01
Record Dates: First submitted 2008-02-25; First posted 2008-03-06 (Estimated); Last update posted 2008-03-06 (Estimated); Status verified 2008-02

CONDITIONS: Hypocalcemia
Keywords: Total thyroidectomy; CND; hypocalcemia; calcium; vitamin D
MeSH Terms: conditions — Hypocalcemia | interventions — Calcium; Vitamin D; Calcium Carbonate; alfacalcidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- C (No Intervention): No supplements after total thyroidectomy and central neck dissection
- D (No Intervention): No central neck dissection group (total thyroidectomy alone)
- A (Active Comparator): Oral calcium plus vitamin D supplements after total thyroidectomy and central neck dissection
  Interventions: Dietary Supplement: Oral calcium plus vitamin D
- B (Active Comparator): Oral calcium alone supplement after total thyroidectomy and central neck dissection
  Interventions: Dietary Supplement: Oral calcium alone

INTERVENTIONS:
Dietary Supplement: Oral calcium plus vitamin D — calcium supplementation took 3 g/day oral calcium (1 g every 8 h) plus 1 mcg/day vitamin D (0.5 mcg every 12 h), beginning on the night of surgery and continuing for 14 days.
  Other Names: calcium carbonate and one-alpha (vitamin D)
  Arms: A
Dietary Supplement: Oral calcium alone — calcium carbonate (3 g/day, 1 g every 8 h)
  Other Names: calcium carbonate (Korea United Pharmaceutical Co, Seoul, Korea)
  Arms: B

SUMMARY:
the increased risk of hypocalcemia following total thyroidectomy plus central neck dissection can be minimized by routine administration of oral calcium and vitamin D supplements during the early postoperative period.

DETAILED DESCRIPTION:
Of patients with differentiated papillary thyroid carcinoma, group D underwent total thyroidectomy alone and groups A-C underwent total thyroidectomy plus CND. The latter were randomized to oral calcium (3 g/day) plus vitamin D (1 mcg/day) (group A, n = 49), calcium alone (group B, n = 49), or no supplements (group C, n = 50). Hypocalcemic symptoms, serum calcium, and parathyroid hormone (PTH) levels were compared among the groups.

ELIGIBILITY:
Inclusion Criteria:

* Differentiated papillary thyroid carcinoma
* Undergoing total thyroidectomy plus central neck dissection

Exclusion Criteria:

* Previous thyroid or neck surgery
* Patients with parathyroid diseases
* Other thyroid malignancies
* Early loss of follow-up without proper evaluation of postoperative serum calcium levels and symptoms

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
The clinical utility of calcium and vitamin D supplements for prevention of hypocalcemia following total thyroidectomy plus central neck dissection | To postoperative 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Lyel Roh, MD, PhD, Principal Investigator — Asan Medical Center & Chungnam National University Hospital
Locations (1):
- Chungnam National University Hospital, Daejeon, South Korea

REFERENCES:
- [Background] Bellantone R, Lombardi CP, Raffaelli M, Boscherini M, Alesina PF, De Crea C, Traini E, Princi P. Is routine supplementation therapy (calcium and vitamin D) useful after total thyroidectomy? Surgery. 2002 Dec;132(6):1109-12; discussion 1112-3. doi: 10.1067/msy.2002.128617. PMID 12490862
- [Result] Moore FD Jr. Oral calcium supplements to enhance early hospital discharge after bilateral surgical treatment of the thyroid gland or exploration of the parathyroid glands. J Am Coll Surg. 1994 Jan;178(1):11-6. PMID 8156110
- [Derived] Roh JL, Park JY, Park CI. Prevention of postoperative hypocalcemia with routine oral calcium and vitamin D supplements in patients with differentiated papillary thyroid carcinoma undergoing total thyroidectomy plus central neck dissection. Cancer. 2009 Jan 15;115(2):251-8. doi: 10.1002/cncr.24027. PMID 19117033